CLINICAL TRIAL: NCT01210820
Title: A Prospective Single Center Study To Evaluate the Feasibility of Intrastromal Arcuate Keratotomy Performed With the IntraLase iFS™ Femtosecond Laser System
Brief Title: Feasibility of iFS™ for Intrastromal Arcuate Keratotomy (ISAK) Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMTO-102-ISAK
Record Dates: First submitted 2010-09-24; First posted 2010-09-29 (Estimated); Results first posted 2013-04-26 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Refractive Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Natural Astigmatism (Experimental): Subjects with refractive astigmatism and no prior history of ophthalmic surgery. May include subjects with cataracts.
  Interventions: Device: iFS™ Femtosecond Laser System
- Post cataract with residual astigmatism (Experimental): Subjects who have had cataract removal surgery but have residual astigmatism.
  Interventions: Device: iFS™ Femtosecond Laser System

INTERVENTIONS:
Device: iFS™ Femtosecond Laser System — intrastromal arcuate cuts made with iFS™ femtosecond laser
  Other Names: iFS™ is part of the product brand name - there is no expanded acronym

SUMMARY:
The results of this trial will demonstrate that ISAK performed with the iFS™ femtosecond laser is a safe procedure.

DETAILED DESCRIPTION:
Surgeon will perform intrastromal arcuate keratotomy in arc segment patterns using the iFS™ femtosecond laser to treat subjects with refractive astigmatism.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, of any race, and at least 21 years of age at the time of the pre-operative examination and signing the consent form
2. Refractive error, no limitation on spherical refractive myopia or hyperopia and refractive astigmatism of 0.75 to 7.00 diopters (D) in the operative eye
3. Best Spectacle Corrected Distance Visual Acuity (BSCVA)

   * Group 1: Natural astigmatism, no cataract: BSCVA of 20/25 or better in both eyes
   * Group 1: Pre cataract surgery, no BSCVA criteria in the operative eye
   * Group 2: Post cataract surgery, BSCVA of 20/25 or better in both eyes
4. Uncorrected Visual Acuity (UCVA) of 20/40 or worse in the operative eye
5. Demonstration of agreement in the operative eye: Corneal astigmatism (as determined by keratometry) must be in agreement with refractive astigmatism (as determined by manifest refractions) as follows: Within ≤ 0.75 D in magnitude and within 15° axis when cylinder ≤ 1.5 D or 10° axis when cylinder > 1.5 D.
6. Preoperative central and peripheral (in planned treatment area) pachymetry of ≥ 500 um in the operative eye
7. Keratometry must be between 38.0 (flat) and 48.0 D (steep) in the operative eye
8. Corneal power (diopters) difference at the 3mm point from topographic center shall be ≤ 1D at the steepest meridian, by topography measurements in the operative eye
9. Intraocular pressure (IOP) of 12 to 21 mm Hg in the operative eye with no glaucomatous retinal changes
10. Stable refractive error in the operative eye, based on an exam (or prescription) at least 6 months prior to the pre-operative examination, and as compared to the pre-operative manifest refraction, must be ≤ 0.75 D (sphere and cylinder) and axis within 15 degrees for eyes with cylinder > 0.5D.
11. Subjects who have worn a contact lens in the operative eye within the past 30 days must remove the soft lens at least 2 weeks prior and a rigid or toric lens at least 3 weeks prior to baseline measurements. In addition, rigid or toric lens wearers must demonstrate stability in topography, keratometry and refraction before proceeding with surgery. Refractive stability is defined as a change of not more than 0.50 D in manifest sphere, cylinder, or keratometry (either axis) as compared to the unadjusted preoperative refraction in two visits at least one week apart.
12. Willing and capable of returning for follow-up examinations for the duration of the study
13. Subject must sign and be given a copy of the written Informed Consent Form

Exclusion Criteria:

1. Abnormal topography, including evidence of keratoconus or pellucid marginal degeneration, in either eye
2. Irregular astigmatism in the operative eye
3. Evidence of clinically significant corneal opacity/scar in the operative eye within an 8 mm diameter zone of the visual axis
4. Women who are pregnant, breast-feeding, or intend to become pregnant over the course of the study, as determined by verbal inquiry
5. Concurrent use of topical or systemic medications that may impair healing, including but not limited to: antimetabolites, isotretinoin (Accutane®) within 6 months of treatment, and amiodarone hydrochloride (Cordarone®) within 12 months of treatment
6. History of any of the following medical conditions, or any other condition that could affect wound healing: collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or herpes simplex, endocrine disorders (including, but not limited to unstable thyroid disorders and diabetes), lupus, and rheumatoid arthritis
7. History of active ophthalmic disease or other non-refractive abnormality (including, but not limited to, corneal dystrophy, symptomatic blepharitis, recurrent corneal erosion, dry eye syndrome, neovascularization > 1mm from limbus), retinal detachment/repair, at risk for developing strabismus, or with evidence of glaucoma or propensity for narrow angle glaucoma NOTE: Subjects with open angle glaucoma, regardless of medication regimen or control, or an IOP greater than 21 mm Hg at baseline, are specifically excluded from eligibility.
8. Known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course
9. Participation in any other conflicting ophthalmic drug or device clinical study during the period of participation in this clinical investigation -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Tarantino, OD, Study Director — Abbott Medical Optics
Locations (1):
- Paracelsus Medizinische Privat-Universitat, PMU, Salzburg, Salzburg, Austria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from an Ophthalmic medical clinic during the period of July 2010 to April 2011.
Groups:
- Natural Astigmatism: Subjects with refractive astigmatism and no prior history of ophthalmic surgery. May include subjects with cataracts.
  iFS™ Femtosecond Laser System : intrastromal arcuate cuts made with iFS™ femtosecond laser
- Post Cataract With Residual Astigmatism: Subjects who have had cataract removal surgery but have residual astigmatism.
  iFS™ Femtosecond Laser System : intrastromal arcuate cuts made with iFS™ femtosecond laser
Period: Overall Study
Arm/Group | Natural Astigmatism | Post Cataract With Residual Astigmatism
Started | 17 | 4
Completed | 17 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Natural Astigmatism: Subjects with refractive astigmatism and no prior history of ophthalmic surgery. May include subjects with cataracts.
  iFS Femtosecond Laser System : intrastromal arcuate cuts made with iFS femtosecond laser
- Post Cataract With Residual Astigmatism: Subjects who have had cataract removal surgery but have residual astigmatism.
  iFS Femtosecond Laser System : intrastromal arcuate cuts made with iFS femtosecond laser
- Total: Total of all reporting groups
Arm/Group | Natural Astigmatism | Post Cataract With Residual Astigmatism | Total
Number analyzed (Participants) | 17 | 4 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (12.4) | 61 (12.1) | 65 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 10 | 1 | 11
Region of Enrollment [Number; unit: participants]
  Austria | 17 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Refractive Astigmatism
Description: Change in mean cylinder (assessed by manifest refraction) compared to baseline.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Diopter of cylinder change
Arm/Group | Natural Astigmatism | Post Cataract With Residual Astigmatism
Number analyzed (Participants) | 17 | 4
Diopter of cylinder change | -0.97 (0.43) | -0.81 (0.35)

2. Primary Outcome: Change in Keratometric Cylinder
Description: Change in mean keratometric cylinder (as measured by keratometry) compared to baseline.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Diopters of astigmatism change
Arm/Group | Natural Astigmatism | Post Cataract With Residual Astigmatism
Number analyzed (Participants) | 17 | 4
Diopters of astigmatism change | -0.81 (0.62) | -0.63 (0.78)

ADVERSE EVENTS:
Arm/Group | Natural Astigmatism | Post Cataract With Residual Astigmatism
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/4
Other Adverse Events (participants affected / at risk) | 0/17 | 0/4

LIMITATIONS AND CAVEATS:
This evaluation was performed on a small number of subjects and should be repeated in a larger number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 1 month prior to any proposed submission for publication or presentation of Trial data or other findings related to the Trial, the Institution will provide the Sponsor with a manuscript for review, comment, and approval. Under no circumstances shall the Institution or PI publish or disclose the Sponsor's confidential Information without the Sponsor's prior written approval.The manner in which the publication will be generated will be negotiated between the Sponsor and PI.